CLINICAL TRIAL: NCT05262309
Title: An Open-label, Randomized, Parallel-arm Study Investigating the Efficacy and Safety of Intravenous Administration of Pamrevlumab Versus Standard of Care in Patients With COVID-19 (FibroCov-01 / FGCL-3019-IST-014)
Brief Title: An Open-label, Randomized, Parallel-arm Study Investigating the Efficacy and Safety of Intravenous Administration of Pamrevlumab Versus Standard of Care in Patients With COVID-19
Acronym: FibroCov-01
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3135
Record Dates: First submitted 2021-06-07; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2021-06

CONDITIONS: COVID-19 Respiratory Infection; COVID-19 Pneumonia; Covid19
MeSH Terms: conditions — COVID-19 | interventions — pamrevlumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pamrevlumab (Experimental)
  Interventions: Drug: Pamrevlumab
- Standard of care (No Intervention)

INTERVENTIONS:
Drug: Pamrevlumab — Pamrevlumab dosing, 30 mg/kg IV, will be administered at day 1, day 7 and day 14.
  Based on Investigator's decision, treatment may be continued every 3 weeks after day 14, up to 11 weeks.
  Arms: Pamrevlumab

SUMMARY:
This is a randomized, open-label, parallel-arm study to investigate the efficacy and safety of pamrevlumab in patients with documented SARS-CoV-2 infection. The study consists of screening, a treatment period, and a follow-up period.

The study will enroll patients who have been hospitalized and who are not currently on invasive mechanical ventilation. The treatment period is open ended, and patients will be randomized to treatment with pamrevlumab or standard of care in a 1:1 ratio according to a pre-generated randomization list. Pamrevlumab dosing, 30 mg/kg IV, will be administered at day 1, day 7 and day 14. Based on Investigator's decision, treatment may be continued every 3 weeks after day 14, up to 11 weeks. A follow-up by visit or phone call will be performed 8 and 12 weeks after the end of the last dose of treatment. The treatment period for an individual patient will not exceed 11 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Documented COVID-19 infection
* Age >=18 to <=80 years
* Interstitial pneumonia (findings of consolidation or ground glass opacities as assessed by chest HRCT)
* Respiratory distress, defined as PaO2/FiO2 ratio of >=100 <=300 mmHg, requiring supplemental oxygen and hospitalization

Exclusion Criteria:

* Invasive mechanical ventilation at screening
* Pregnancy
* Incapacity to express a valid informed consent
* Known hypersensitivity to monoclonal antibodies used as experimental drugs for any clinical indication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients not on ventilatory support | 15 days

SECONDARY OUTCOMES:
PaO2/FiO2 ratio as categorical variable | Day14
For patients already on mechanical ventilator at time of randomization, the number of days on ventilator after randomization. | up to 12 weeks
For patients not on mechanical ventilator at time of randomization, the number of days not requiring invasive mechanical ventilation | up to 12 weeks
PaO2/FiO2 ratio as continuous variable | Day14
Resting SpO2 adjusted by FiO2 | Day14
Change in oxygen supplementation requirements (liters per minute) | Day14
Quantitative and qualitative assessment of pulmonary lesions by chest HRCT scans at baseline and at day 14 and week 12 | Day 14 and week 12
Time to hospital discharge | up to 12 weeks
Time to all-cause mortality | up to 28 days
Proportion of patients discharged from ICU and alive | within 28 days
Proportion of patients alive | within 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, Rome, Roma, Italy

REFERENCES:
- [Derived] Sgalla G, Leone PM, Gualano G, Simonetti J, Comes A, Verdirosi D, Di Gennaro F, Larici AR, Ianniello S, Cicchetti G, Fusco N, Pani M, Palmieri F, Richeldi L. A randomized trial of pamrevlumab in patients with COVID-19 pneumonia. Respirology. 2023 Oct;28(10):954-957. doi: 10.1111/resp.14575. Epub 2023 Aug 21. No abstract available. PMID 37605035